CLINICAL TRIAL: NCT04528537
Title: Adaptation and Validation of the Quality of Recovery 15-questionnaire for the Postanesthesia Care Unit
Brief Title: Validation of the Quality of Recovery Questionnaire for the Postanesthesia Care Unit (QoR-PACU)
Status: Completed | Type: Observational
Sponsor: Marlene Fischer (Other)
Responsible Party: Sponsor-Investigator, Marlene Fischer, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Other Study IDs: PACQoR3
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Quality of Recovery in the Postanesthesia Care Unit
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — 16-item quality of recovery questionnaire for the postanesthesia care unit (QoR-PACU)

SUMMARY:
Quality of recovery after surgery and anesthesia is an important endpoint in perioperative medicine. Several questionnaires have been developed that assess the patient's perception on postoperative recovery at 24 h after surgery. This study aims to adapt validate the Quality of Recovery 15-questionnaire for application in the postanesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* general anesthesia
* fluency in German

Exclusion Criteria:

* postoperative intensive care unit stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-cardiac surgery under general anesthesia in a postanesthesia care unit at a tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
16-item quality of recovery questionnaire for the postanesthesia care unit (QoR-PACU) | up to 4 hours following extubation
  Validity of the QoR-PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No